Pilot Testing a Home-Based Rehabilitation Intervention Designed to Improve Outcomes of Frail Veterans Following Cardiothoracic Surgery

NCT03299101

7/24/2020

#### 1.0 \* Study Name:

Home-based Rehabilitation Before Cardiothoracic Surgery (Pilot)

# 2.0 \* Brief Description (using layman's terms) - 500 words or less:

Frail Veterans are at increased risk for poor surgical outcomes, and as the Veteran population grows older and more frail, there is a critical need to identify effective strategies for reducing surgical risks for these patients. Prior research shows that inter-disciplinary rehabilitation strategies deployed after surgery enhance recovery and improve outcomes by building strength and improving nutrition. We believe that similar improvements may be obtained by using similar interventions before surgery to "prehabilitate" patients' capacity to tolerate the stress of surgery. The proposed research will examine the feasibility of a novel, multifaceted, home-based prehabilitation intervention designed to improve functional capacity and postoperative outcomes for frail Veterans anticipating cardiothoracic surgery. Findings from the study will inform the design of a larger randomized controlled trial of the prehabilitation intervention. If proven effective, prehabilitation could benefit as many as 42,000 frail Veterans who are scheduled for major elective surgery each year.

## \* Abstract. Please provide a brief description of the study.

Background: Frail Veterans are at increased risk for poor surgical outcomes. Although surgical techniques have advanced to a level where surgery on very old adults is feasible, if a patient is also frail, the stress of surgery may overwhelm their adaptive capacities, placing them at increased risk of mortality, morbidity, and institutionalization even if surgery is technically successful. Frailty is a clinical syndrome that is commonly characterized by muscle atrophy, diminished strength and speed, decreased physical activity, and exhaustion. It is independent of any specific disease, but it increases with age and worsens disease prognoses by diminishing capacity to tolerate stressors. Thus, while surgery is often indicated for older patients, frail candidates are less likely than robust counterparts to tolerate the procedure and/or recover functional capacity. In fact, recent VA data demonstrate that frailty is a more powerful predictor of increased perioperative mortality, morbidity, length of stay, and cost than predictions based on age or comorbidity alone. As the Veteran and US populations grow older, frailty will increase, making it critically important to identify effective strategies for improving the surgical recovery and outcomes of frail patients.

"Prehabilitation" has the potential to improve surgical outcomes among the frail. Prior research demonstrates that inter-disciplinary rehabilitation strategies deployed after surgery enhance recovery and improve outcomes by building strength and improving nutrition. Based on this success, there is growing interest in "prehabilitation", which is a similar intervention deployed before surgery. By modifying physiological and environmental risks, prehabilitation aims to augment patients' capacity to compensate for the stress of surgery itself and the convalescent period thereafter. Frail patients may benefit disproportionately from prehabilitation because they have diminished capacity to endure the procedure and/or recovery. Preliminary evidence suggests that preoperative exercise interventions improve surgical outcomes. However, prehabilitation has not yet been studied in either Veteran or specifically frail populations, and no prior studies used home-based prehabilitation strategies to safely minimize travel-related barriers to participation.

Objectives: We will examine the feasibility of a novel, multifaceted, home-based prehabilitation intervention designed to improve functional capacity and postoperative outcomes for frail Veterans anticipating cardiothoracic surgery. Specific aims are to:

- (1) Estimate rates of recruitment, retention, and adherence to the intervention; and evaluate participation barriers.
- (2) Measure changes over time in frailty, physical function, pulmonary function, nutrition, and health-related quality of life at baseline, the day of surgery, and 30 and 90 days after surgery.
- (3) Explore changes in postoperative mortality, major complications, length of hospital stay, and level of independent living using case-matched historical controls.

Methods: This single-arm pilot study will enroll a consecutive cohort of up to 50 Veterans identified as frail using a standardized frailty assessment and scheduled for major cardiothoracic surgery at the VA Pittsburgh Healthcare System. The 4 week long prehabilitation regimen will include: (a) aerobic conditioning, (b) strength and coordination training, (c) respiratory muscle training, and (d) nutritional coaching and supplementation. Pre- and post-prehabilitation assessments will include: (a) frailty; (b) physical function; (c) pulmonary function; (d) nutrition; and (e) health-related quality of life. Postoperative outcomes will include length of stay, mortality

Research Study Methods

View: 4 Research study methods

\* Research Procedures/Interventions:

#### **Research Procedures/Interventions:**

- **C.1. Overview.** In this single-arm pilot study, we will enroll a consecutive cohort of up to 50 Veterans identified as frail using a standardized frailty assessment and scheduled for major cardiothoracic surgery at the VA Pittsburgh Healthcare System. The 3-6 week long prehabilitation regimen will include: (a) aerobic conditioning, (b) strength and coordination training, (c) respiratory muscle training, and (d) nutritional coaching and supplementation. Pre- and post-prehabilitation assessments will include: (a) frailty; (b) physical function; (c) pulmonary function; (d) nutrition; and (e) health-related quality of life. Using physical performance tests, biomarkers, chart review, survey instruments, and patient logs, we will assess the feasibility of the recruitment, randomization, retention and assessment procedures, compensating patients for their time. Prehabilitation will not last more than 4 weeks for CABG patients. However, for non-cardiac thoracic patients, prehabilitation may be extended out to 6 weeks if the surgeon and patient so choose.
- C.2. Eligibility criteria. We will recruit frail patients (i.e., RAl≥16 and Physician /Provider request for patient with RAI<16) scheduled for a CABG or Valve Surgery. Major non-cardiac thoracic surgery is defined according to VA Surgical Quality Improvement Program (VASQIP) criteria that include cases requiring general, epidural, or spinal anesthesia. It includes 193 unique CPT codes ranked by complexity (26 standard, 146 intermediate, and 21 complex) and excludes 58 low risk "minor" surgical procedures with limited morbidity (e.g., bronchoscopy, percutaneous lung biopsy). From these major surgeries, we will include those procedures that deliberately violate the visceral or parietal pleura with something larger than an 18 gauge needle. For example, we will include lung and esophagus resections of all kinds, but exclude thoracentesis. Exclusion criteria are designed to ensure participant safety in prehabilitation exercises (e.g., low-risk, stable cardiac disease without significant symptoms, arrhythmias, hemodynamic instability or critical coronary lesions). Based on historical data, we expect 2/3<sup>rds</sup> of eligible

patients to exhibit mild frailty (RAI 16-25) with essentially intact independence and capacity for prehabilitation. Higher degrees of frailty may impose barriers to full participation, but characterizing those limitations is an important component of this pilot. We will stratify enrollment to ensure approximately equal enrollment of cardiac and non-cardiac thoracic patients.

- **C.3. Prehabilitation procedures.** Prehabilitation will last 3-6 weeks—a time frame that does not delay surgery, corresponds to the typical lag for surgical scheduling, and strikes a pragmatic balance between improving physiologic reserve without unduly delaying definitive surgical therapy. Although the training intervention is only 3-6 weeks, studies repeatedly demonstrate neuromuscular strengthening, adminished inflammation, and respiratory improvements within this time. Further, the program also fosters continuity between preoperative training and traditional postoperative rehabilitation, facilitating rapid mobilization and progressive exercise after surgery. Strategies like this enhance functional recovery and reduce the risks of subsequent episodes of disability (e.g., readmission or loss of independence). S8.78-81 If clinical contexts such as neoadjuvant chemotherapy or worsening angina require shorter (or permit longer) durations of training, we will examine these events in order to inform the optimal duration of prehabilitation for a larger clinical trial.
- (a) Safety. Prehabilitation will begin in a telemetry-monitored, hospital-based setting to train patients in the home-based exercises and establish safe targets of exertion. If and as safety is established, exercise will shift to the home with weekly telephone/ VA Video Connect contact to ensure safety and reinforce technique. Remote telephone and VA Video Connect monitoring will be enhanced by the relationships, familiarity, and trust established during the hospital-based sessions. Although safety concerns will require some patients to complete all exercise in monitored, hospital-based settings, we anticipate that many patients will safely transition to home-based exercise after 1-4 hospital-based sessions. Study staff will initiate withdrawal procedures for patients who demonstrate insufficient cognitive or physical capacity to safely carry out the prescribed activities.
- (b) Hospital-based training. Twice weekly 1-hour hospital sessions will be closely monitored and continue until participants demonstrate: (a) mastery of prehabilitation techniques; and (b) compliance with safe targets of exertion that do not induce cardiac symptoms. All patients will complete at least 1 sessions with telemetry to rule-out significant arrhythmia, but they will continue as long as needed to ensure that exercise can safely shift to the home. Aerobic training will focus on seated pedaling. Leg pedaling is preferred, but in cases of lower extremity disability, upper extremity exercise will be implemented. After a 3-5 minute warm-up at a low intensity of an 7-9 on the Borg Rating of Perceived Exertion (RPE) scale, 22 patients will be coached to reach 30 minutes of continuous (through bouts of 10 minutes or more to work up to the 30minutes), moderate exertion (RPE 11-13). If this exertion induces cardiac symptoms, the target will be adjusted down until a safe level is established. Strength training will use body weight and resistance bands (TheraBand™) at RPE 11-13 to focus on a spectrum of antagonist muscles to support the core abdominal and thoracic muscles impacted by surgery. Coordination training will involve exercises designed to strengthen the proper form of transitional movements required after surgery such as lying-to-side-lying, side lying-to-sitting, seated scooting, and sitting-to-standing. Respiratory muscle training (RMT) requires that subjects inspire and exhale through a mouthpiece at a comfortable rate using diaphragmatic breathing techniques while wearing a nose clip. The RMT device prohibits subjects from inhaling or exhaling until specific negative or positive pressures are achieved. Thresholds devices will be used and set at 40% of each patient's maximal inspiratory pressure (MIP) performed on the Pro2 device. Training will involve 5-20 breaths depending on patients capacity on the threshold device with resistance increased weekly based on RPE with a goal of moderate exertion (RPE 11-12) on both inhalation and exhalation.

- (c) Home-based Training. Home-based training will increase gradually to reach the goal duration of 60 minutes allocated between strength training 3 days/week and aerobic, RMT and coordination training 5 days/week. Each session will begin with warm up before focused aerobic (pedal exerciser), strength, coordination, and RMT training, followed by cool down and stretching that matches the routines established during hospital-based training. Each patient will be given a portable, folding pedal exerciser that can be placed on the floor for leg pedaling or on a table for arm pedaling. Based on methods that successfully transition cardiac rehabilitation to the home, <sup>2</sup> exercise physiologists will use weekly, remote, telephone-based/ VA Video Connect calls to maintain relationship, answer questions, adjust goals and coach patients regarding their personally tailored prehabilitation regimens. Patients will record details of each training session in log books, and they may return to the hospital biweekly to assess progress in physical performance, or their biweekly session may be completed via VA Video Connect, at which time exercise physiologists will (a) adjust training goals and exercises, (b) remediate technique as needed; and (c) assess the safety of continued home exercise. Family members or other caregivers can assist patients in completing the log books if needed. Training regimens such as these have been shown to be both safe and effective among the frail elderly.<sup>83</sup>
- (d) Nutritional Counseling. Standard or care consults with the VAPHS Nutrition Services will coincide with the initial IMPACT clinic visit. Staff nutritionists will administer the Subjective Global Assessment (SGA) of nutrition to identify nutritional needs and classify the patient as either normal or mildly, moderately or severely malnourished. All patients will receive best practice nutritional counseling focused on lean, high protein foods in preparation for surgery. Cardiac rehabilitation personnel/research staff will be trained to assess and reinforce progress on these dietary practices. In addition, standard of care nutritional supplementation will be prescribed to malnourished patients, including Impact® Advanced Recovery, an immunomodulating formula shown to improve outcomes after major surgery. Supplements will be delivered to patient's homes. Patients will also record their meals and supplements in log books, and cardiac rehab personnel/research staff will be trained to monitor and encourage consumption of the supplements as prescribed during the hospital-based coaching sessions. Family members or other caregivers can assist patients in completing the log books if needed.
- **(e)** Occupational and Physical Therapy (OT/PT). We will arrange for a standard OT/PT consult to coincide with either the initial IMPACT clinic visit or the first scheduled visit to the Cardiac Rehabilitation facility. Staff therapists will perform routine, standardized assessments of the patient's home, environment and mobility, prescribing and supplying indicated durable medical equipment to aid mobility, exercise, and safe transition to independent living at home after the proposed surgery. As per their usual protocol, the PT/OT consult will consult with the Social Work services to adequately assess the home environment and supports in anticipation of postoperative discharge planning.
- **C.4. Assessment Schedule (Table1).** As shown in Table 1, research staff will collect baseline data, including demographics, living location, physical performance, and nutrition, at the time of recruitment. Assessments will continue every 2 weeks up to and including the day of surgery, and then postoperatively at 30 and 90 days. Even among the robust, physical performance deteriorates immediately after surgery, but returns to baseline by 90 days. Among the frail, the deterioration may endure, increasing the severity of frailty. Physical Performance Tests will be administered by exercise physiologists in the VAPHS Rehabilitation facility, located near the IMPACT clinic, and thus convenient for patients. Nutrition Assessments include serum prealbumin and c-reactive protein collected each time the participation is onsite for an assessment by a hospital phlebotomists, and the 7-point SGA administered by hospital nutritionists at baseline and again on the day of surgery. Patient Logs will assess patient adherence with the prehabilitation regimen and document progress. Family members or

other caregivers can assist patients in completing the log books if needed. <u>Survey Instruments</u> will be administered either face to face, by telephone/ VA Video Connect, or by mail, depending on patient preference. Responses will be entered directly into REDCap using a project utility distinct from the RAI measurement tool. For patients electing surveys by mail, we will send printed copies of the Redcap forms with a self-addressed, stamped envelope for return. Responses on returned surveys will be keyed into Redcap before storing the paper surveys in locked cabinets. <u>Chart reviews</u> will be completed by research staff to determine details of the surgical procedure, postoperative mortality, length of stay, and major complications. <u>Patient Interviews</u> will be conducted to evaluate barriers to prehabilitation and explore possible solutions. We will also track the time required to complete each measure to inform the design of the subsequent multi-center trial.

Assessments will end after the assessment planned for 90 days after the surgery. Ideally, patients will return to the hospital for this final visit to conduct measures of physical performance and nutrition along with the survey instruments. However, if they are unable to make the visit, we will conduct the surveys over the phone.

Minimizing the Burden of Assessments: Some participants in this study will be concurrently enrolled in a related study of frailty and preoperative palliative care consultation (Pro1840). Some of the outcome assessments planned for Pro 1840 are identical to those planned here. When a participant is enrolled in both studies (Pro1840 and Pro 2192) the study coordinators will work together to ensure that participants do not have to complete identical assessments twice. At any given time point when potentially duplicative assessments could occur, study staff will record the participant's singular response to a duplicative question simultaneously into the case report forms (CRFs) of each separate study. This could be accomplished by having a two separate study staff on the phone or in the room as the patient is interviewed. It could also be accomplished by having a single cross-listed staff member (e.g., listed on the staff form of both studies) administer the assessment and record the responses into the separate CRFs of each study at the same sitting. Additionally, some participants may be concurrently enrolled in a minimal risk study (PI James Ibinson MD; Pro1843) that has similar inclusion criteria. However participation in Pro1843 will not impact the outcomes of this protocol (2192).

To reduce patient burden due to travel once a patient has been determined to be safe to take part in home exercise they will have the option to complete an remote biweekly assessment via VA VideoC onnect. Biweekly Assessments for patients that are unable to make it to the hospital will complete an remote, home-based biweekly assessment while on VA Video Connect with research staff members. VA Video Connect will be used in conjunction with Bluetooth connected peripheral monitors that record and transmit blood pressure, pulse, and oxygen saturation in real time. Single lead cardiac telemetry will also be used once this peripheral is made available (date pending). We will also monitor the patient visually through the video feed to ensure safety. The remote assessment will included the following items form the standard assessment: Five chair rises (standing and siting form a chair 5 times), two 4 meter walks at usual walking speed, assessment of breathing capacity on the threshold trainer (adjusted by RPE scale with goal of RPE 11-13), and if space allows a modified 6 minute walk test.

| Table 1: Assessment Schedule | | | | | |
|---|---|---|---|---|---|
| | Baseline | Every other<br>Week | Day of | 30 Days | 90 Days |
| | | In-hospital | surgery | post-op | post-op |
| Demographics | | | | | |
| Age, sex, race, ethnicity, etc | Х | | | | |
| Procedure-related variables | Х | | | Х | |
| Living Location | Х | | Х | Х | Х |
| Physical Performance | | | | | |
| SPPB | Х | X | Х | | х |
| MIP & MEP | Х | X | Х | | х |
| 6 Minute Walk Test | Х | Х | Х | | Х |
| Frailty (multiple measures) | Х | X | Х | | х |
| Nutrition | | | | | |
| Prealbumin (biweekly) | Х | X | Х | | х |
| вмі | Х | X | Х | | х |
| Subjective | X | | Х | | |
| Global Assessment | ^ | | ^ | | X |
| Compliance | | | | | |
| Patient Logs | | X | Χ | | |
| Barrier Assessment | X | X | Χ | X | X |
| Outcomes | | | | | |
| Mortality | | | | X | Х |
| Length of Stay | | | | X | |
| Major Complications (30 day) | | | | Х | |
| Quality of Life | Х | | Х | | Х |
| Quality of Surgical Care (Pre) | | | Х | | |
| Quality of Surgical Care (Post) | | | | Х | |
| Measure of Flourishing | Х | | X | | Х |
| Measures of Decision Quality | Х | | Х | X | Х |

### C.5. Variables Assessed.

- Age, sex, race, ethnicity and socioeconomic status will be assessed by direct patient survey or chart review.
- <u>Procedure-related variables</u> will include the CPT codes of the initially planned operation as well as the
  operation actually performed. We will also abstract from the chart the type of anesthesia, the duration
  of the procedure, and the disposition of the patient at the end of surgery (e.g., discharge v. admission)
- <u>Living Location</u> is the environment where patients are living before and after the index operation (i.e., home, nursing home, etc). It will be assessed by direct patient survey or chart review and followed as an outcome.
- Short Physical Performance Battery (SPPB) is a test of balance, gait, strength, and endurance that combines gait speed, repeated chair stands and balance tests that together take less than 5 minutes to complete. Each of the 3 tests are scored on a scale from 0-4 with a combined score ranging from 0-12

with lower scores indicating worse performance. <sup>26</sup> Scores below 8 or 10 are interpreted as poor performance. <sup>82</sup> The SPPB accurately predicts adverse outcomes such as disability, hospitalization, nursing home admission, frailty and mortality, and is becoming the reference standard in rehabilitation literature. <sup>82-86</sup>

- <u>6 Minute Walk Test</u> is a standard measure of physical performance that measures the total distance traversed in 6 minutes, measured in meters. Clinically significant differences can be quantified in as little as 30 meters. This is an exploratory measure that will only be administered if time allows. As a pilot study, we aim to determine what kinds of assessments are feasible in this group.
- Maximal Inspiratory & Expiratory Pressures (MIP & MEP) are the standard metrics of respiratory muscle strength<sup>27</sup> and will be measured using the TIRE device described above (D.6c). It has been shown that changes as small as 15 cm  $H_2O$  can significantly reduce postoperative pulmonary complications and length of stay.<sup>78</sup>
- Frailty will be assessed through several measures because no single measure of frailty captures the breadth of the syndrome. In addition to the RAI described above, we will quantify the Hopkins & Edmonton Frail Scales and independently analyze the gait speed and handgrip strength that is part of the Hopkins Frail Scale. We recently developed a streamlined approach to measuring all of these metrics simultaneously in a parsimonious exercise that takes <5 minutes to administer.</p>
- Hopkins Frail Scale encompasses slowness, weakness, weight loss, low physical activity, and exhaustion with ≥3/5 criteria required to distinguish frailty.<sup>31,32</sup> It is the most frequently cited tool shown to predict mortality and disability in large cohorts of community-dwelling elders and surgical patients.
- Edmonton Frail Scale is an 11-item survey that assesses 8 dimensions of frailty. Each item is scored 0, 1, or 2 with higher scores indicating greater frailty. The total score ranges from 0-17 with good inter-rater reliability (k = 0.77), moderate internal consistency (alpha=0.62), and strong correlation with a geriatrician's assessment of frailty (r=.64, p<.001).88</p>
- <u>Gait speed</u> is one key measure of frailty<sup>76,97,98</sup> that has excellent inter-rater reliability (intraclass coefficient 0.88-0.96) and test-retest reliability (intraclass coefficient 0.86-0.91).
- <u>Handgrip Strength</u> has also been demonstrated to have key utility as an index of frailty. 32,89 A grip dynamometer will be used, averaging 2 serial assessments from the dominant hand.
- Prealbumin will be measured with standard serological testing. Changes can be detected in days, and it is the best available biomarker of nutrition.<sup>90,91</sup> However, because prealbumin can function as an acute phase reactant, we will also concurrently measure c-reactive protein as a measure of inflammation and interpret prealbumin as proposed by Jensen, et al.<sup>92,93</sup>
- Body Mass Index (BMI) will be calculated from height and weight assessed each week at the Cardiac Rehab facility, and is considered the most suitable, objective anthropometric indicator of nutritional status,<sup>94</sup> and changes in BMI have been shown to predict survival in the elderly.<sup>95</sup>
- Subjective Global Assessment of Nutrition (SGA) is the standard approach to nutritional assessment.<sup>96</sup> It evaluates multiple domains of nutrition and reliably categorizes patients into 1 of 4 categories: normal, mild-, moderate- and severely malnourished. We will use the 7-point SGA (See Appendix) because it is sensitive to 1-point changes in as little as 1 month and has excellent inter-rater reliability (k=.726).<sup>28</sup>
- Compliance with Prehabilitation. Each patient will receive a prehabilitation log book in which they will record details about their home-based regimen, including the date of training, duration and intensity of exercise, IMT repetitions and threshold pressures, nutritional supplements consumed, dietary intake, and pedometer data (e.g., step counts at the beginning and end of each training session). They will be coached in the use of this log at each hospital session. Data from the logbook will be collected from patients weekly and entered into the database for analysis. In addition, because the pedometer stores 7 days of data, and the exercise physiologists will record daily step counts as a measure of overall activity at each hospital session.

- <u>Barrier Assessment</u> will be conducted through face-to-face or telephone interviews with participants who encounter difficulty with recruitment to, retention in, or adherence with the training regimens. Barriers, including advanced frailty and cognitive deterioration will be described and participants will be asked to propose facilitators that might remove or minimize the barrier in future. Interviews will not be elaborate, but the questions are detailed in the case report forms. No formal qualitative analysis will be conducted, but responses will be collated and summarized by research staff. We will not record responses or attempt to create verbatim transcripts, but instead, the research staff conducting the interviews will summarize patient responses and record those summaries in the case report forms.
- <u>Health-Related Quality of Life</u> will be measured with the Assessment of Quality of Life (AQoL-6D) that includes 20 items on a Guttman scale assessing 6 domains: independent living, mental health, relationships, senses, pain and coping.<sup>97</sup> The utility score ranges from -.04 (state worse than death) to 1.0 (full health). It is sensitive to change with a minimum clinically important difference (MCID) of 0.06.<sup>98</sup>
- Quality of Surgical Care will be measured with the Surgical Care Survey (SCS) that includes subscales for quality of pre-surgical care (11 items), day of surgery (6 items), and postoperative care (12 items).
- Flourishing will be measured by the "Secure Flourish" measure, which is 12 items assessing 6 domains: happiness & life satisfaction, mental & physical health, meaning & purpose, character & virtue, close social relationships, and financial & material stability. All items are scored from 0 to 10. This measure is calculating by summing the scores of all six domains.
- Measures of Decision Quality include Decision Regret (5 items), Patient Centeredness of Care (12 items),
   Satisfaction with the Process of Decision Making (14 items), Satisfaction with the IMPACT clinic (8
   items), Satisfaction with the frailty diagnosis (8 items), satisfaction with the palliative care consult (8
   items), and Satisfaction with the surgeon (8 items).
- Mortality. Patients completing the 30- and 90-day surveys will be confirmed alive. For all others, chart
  review including telephone contact with identified surrogates will confirm vital status and date of death
  (if deceased).
- <u>Length of Stay</u> will be calculated from the date of surgery to the date of discharge or transfer from the hospital. We will also record the time spent in the intensive care unit. Intervals will be calculated in days.
- Major Complications will be abstracted from the chart according to VASQIP coding rules (Appendix). The presence or absence of each complication will be recorded separately, but analysis will focus on a dichotomous outcome indicating the occurrence of serious, Clavien-Dindo level IV complications. These include deep wound infections, organ space infections, wound disruption, pneumonia, unplanned intubation, pulmonary embolism, mechanical ventilation for >48 hours, progressive renal insufficiency, acute renal failure, stroke, coma, cardiac arrest, myocardial infarction, bleeding in excess of 4 units, deep vein thrombosis, sepsis and C. difficile colitis. This approach to analyzing complications has been shown to correlate with frailty. Co-I and Chief of Surgery Mark Wilson has authorized the VASQIP nurse abstractor to use standard VASQIP procedures to code the charts of participating patients.

<u>Incidental Findings:</u> If any of these tests generate an incidental finding of sufficient clinical significance to warrant review by the patient's primary care physician (PCP), we send the test results to the PCP and follow up with an encrypted email. We will also telephone the patient within a week to inform the patient of the finding and the planned PCP follow-up.

C.8. Data Analysis will focus on the feasibility of both the intervention and the outcome assessments. 1

(a) General approach for quantitative data. We will first explore the data using descriptive statistics (e.g., means, standard deviations, percentiles, ranges) and graphical techniques (e.g., histograms,

scatter plots) to examine key variables to assess distributional assumptions, the existence of outliers and data sparseness. We will try to minimize the amount of data missing due to dropouts, but will use multiple imputation if indicated.

- (b) Assess the feasibility of a novel prehabilitation intervention by estimating rates of recruitment, retention, and adherence to the intervention, and by evaluating barriers to participation [Aim 1]. We will summarize the total number of eligible patients approached, recruited, and retained through the completion of study procedures 90 days postoperatively, estimating proportions as well as associated confidence intervals (CIs). We will then estimate rates of adherence to the prehabilitation intervention, computing overall and exercise-specific rates (and CIs) for the home and hospital portions of the regimen. Finally, we will qualitatively analyze reported barriers to participation with an eye to identifying potential solutions.
- (c) Ascertain the feasibility of measuring changes over time in frailty, physical function, pulmonary function, nutrition, and health-related quality of life at baseline, the day of surgery, and 30 and 90 days after surgery [Aim 2]. We will summarize the time required to complete each assessment as well as the completeness of data, estimating completion rates with Cls. Graphical analyses will assess simple changes in frailty, physical performance, pulmonary function, nutrition and quality of life over the study period. Although sample size will limit model fit, we will prepare analyses for the larger trial by developing simple mixed models to explore changes over time (baseline and every other week up to the day of surgery, and then 30 and 90 days after). Separate models for each outcome will assess changes, including a fixed effect for time and a random effect for subject. The type of mixed model will depend on the outcome variable with linear mixed models for continuous variables (e.g., RAI, SPPB, 6MWT, MIP, MEP, etc) and generalized mixed models for ordinal/categorical variables (e.g., SGA, frailty phenotype). We will also explore dose-response relationships based on the actual duration of and adherence to the training regimen.
- (d) Explore changes in postoperative mortality, major complications, length of hospital stay, and level of independent living using case-matched historical controls [Exploratory Aim]. We will match each participant to an historical control using local VASQIP data. VASQIP data include variables sufficient to calculate the RAI as well as details about the patient's procedure, comorbidities, outcomes, and a highly reliable prediction of postoperative 30-day mortality. Each historical control will be chosen from VAPHS VASQIP data from the 2 years prior to the study start and matched to the enrolled participant based on procedure, age, RAI score, and VASQIP predicted mortality. We will summarize separately the total number of deaths and major complications at 30 and 90 days for all patients, estimating proportions with associated CIs for the intervention and historical control groups. We will also compute summary statistics (mean, median, standard deviation, range) for length of hospital stay and return to independent living. We will then attempt to assess if differences exist between the groups with regard to these post-operative measures.
- (e) Additional exploratory analyses. Two related pilot studies conducted by the PI use methods similar to those described here (e.g., Pro 1840 & Pro 1754). In particular, these studies collect identical patient reported survey measures and identical physical performance measures. Each study describes analyses of these data to generate reliable estimates of central tendency and dispersion for use in designing future studies. And in the case of this study and Pro 1754, they describe measuring change over time during the pre and post operative period. However, each study has struggled with recruitment leading to smaller than expected sample sizes. Therefore, we plan to transfer de-identified data from Pro 1840 and Pro 1754 into this study to augment the sample size and thereby increase the precision and power

of our estimates. We do not plan or expect data analysis of this augmented sample to differ in any way from that described in 1840 and 1754 and to which the participants gave consent; the only difference is that the value of each participant's data is augmented by joining it to other similar data.

**Please provide a list of references** (Multi-site protocols: You may reference the page numbers in the original protocol):

- 1. Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. May 2011;45(5):626-629.
- 2. Kraemer HC, Mintz J, Noda A, et al. Caution regarding the use of pilot studies to guide power calculations for study proposals. Achives of General Psychiatry. 2006;63:484-489.
- 3. Buckingham SA, Taylor RS, Jolly K, et al. Home-based versus centre-based cardiac rehabilitation: abridged Cochrane systematic review and meta-analysis. Open Heart. 2016;3(2):e000463.
- 4. Taylor RS, Dalal H, Jolly K, et al. Home-based versus centre-based cardiac rehabilitation. The Cochrane database of systematic reviews. Jan 20 2010(1):CD007130.
- 5. Taylor RS, Dalal H, Jolly K, et al. Home-based versus centre-based cardiac rehabilitation. The Cochrane database of systematic reviews. Aug 18 2015(8):CD007130.
- 6. Dalal HM, Zawada A, Jolly K, et al. Home based versus centre based cardiac rehabilitation: Cochrane systematic review and meta-analysis. BMJ. Jan 19 2010;340:b5631.
- 7. Wakefield B, Drwal K, Scherubel M, et al. Feasibility and effectiveness of remote, telephone-based delivery of cardiac rehabilitation. Telemed J E Health. Jan 2014;20(1):32-38.
- 8. Mans CM, Reeve JC, Elkins MR. Postoperative outcomes following preoperative inspiratory muscle training in patients undergoing cardiothoracic or upper abdominal surgery: a systematic review and meta analysis. Clinical rehabilitation. May 2015;29(5):426-438.
- 9. Anderson GS, Deluigi F, Belli G, et al. Training for improved neuro-muscular control of balance in middle aged females. J Bodyw Mov Ther. Jan 2016;20(1):10-18.
- 10. Schoenrath F, Markendorf S, Brauchlin AE, et al. Robot-assisted training for heart failure patients a small pilot study. Acta Cardiol. Dec 2015;70(6):665-671.
- 11. Robert CM, Sean MB. Physiological Reserve and Frailty in Critical Illness. Oxford, UK: Oxford University Press; 2014.
- 12. Walston J, Hadley EC, Ferrucci L, et al. Research agenda for frailty in older adults: toward a better understanding of physiology and etiology: summary from the American Geriatrics Society/National Institute on Aging Research Conference on Frailty in Older Adults. J Am Geriatr Soc. Jun 2006;54(6):991-1001.
- 13. Partridge JS, Harari D, Dhesi JK. Frailty in the older surgical patient: a review. Age and ageing. Mar 2012;41(2):142-147.
- 14. Chen X, Mao G, Leng SX. Frailty syndrome: an overview. Clinical Interventions in Aging. 03/19 2014;9:433-441.
- 15. Afilalo J, Alexander KP, Mack MJ, et al. Frailty assessment in the cardiovascular care of older adults. J Am Coll Cardiol. Mar 4 2014;63(8):747-762.
- 16. Forman DE, Alexander KP. Frailty: A Vital Sign for Older Adults With Cardiovascular Disease. Can J Cardiol. Jun 2 2016.
- 17. Robinson TN, Wu DS, Pointer L, et al. Simple frailty score predicts postoperative complications across surgical specialties. Am J Surg. Oct 2013;206(4):544-550.
- 18. Robinson TN, Wu DS, Stiegmann GV, et al. Frailty predicts increased hospital and six-month healthcare cost following colorectal surgery in older adults. Am J Surg. Nov 2011;202(5):511-514.
- 19. Adams P, Ghanem T, Stachler R, et al. Frailty as a predictor of morbidity and mortality in inpatient head and neck surgery. JAMA otolaryngology-- head & neck surgery. Aug 1 2013;139(8):783-789.
- 20. Makary MA, Segev DL, Pronovost PJ, et al. Frailty as a predictor of surgical outcomes in older

patients. J Am Coll Surg. Jun 2010;210(6):901-908.

- 21. Robinson TN, Wallace JI, Wu DS, et al. Accumulated frailty characteristics predict postoperative discharge institutionalization in the geriatric patient. J Am Coll Surg. Jul 2011;213(1):37-42; discussion 42-34.
- 22. McAdams-DeMarco MA, Law A, Salter ML, et al. Frailty and early hospital readmission after kidney transplantation. American journal of transplantation: official journal of the American Society of Transplantation and the American Society of Transplant Surgeons. Aug 2013;13(8):2091-2095.
- 23. Anderson L, Taylor RS. Cardiac rehabilitation for people with heart disease: an overview of Cochrane systematic reviews. Cochrane Database of Systematic Reviews. 2014(12).
- 24. Handoll HHG, Cameron ID, Mak JCS, et al. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database of Systematic Reviews. 2009(4).
- 25. Hoogeboom TJ, Dronkers JJ, Hulzebos EHJ, et al. Merits of exercise therapy before and after major surgery. Current Opinion in Anaesthesiology. 03/06 2014;27(2):161-166.
- 26. Oosterhuis T, Costa LOP, Maher CG, et al. Rehabilitation after lumbar disc surgery. Cochrane Database of Systematic Reviews. 2014(3).
- 27. Spruit MA. Pulmonary rehabilitation. Eur Respir Rev. Mar 1 2014;23(131):55-63.
- 28. Pouwels S, Stokmans RA, Willigendael EM, et al. Preoperative exercise therapy for elective major abdominal surgery: a systematic review. Int J Surg. 2014;12(2):134-140.
- 29. Cabilan CJ, Hines S, Munday J. The effectiveness of prehabilitation or preoperative exercise for surgical patients: a systematic review. JBI Database System Rev Implement Rep. 2015;13(1):146-187.
- 30. Dunne DF, Jack S, Jones RP, et al. Randomized clinical trial of prehabilitation before planned liver resection. Br J Surg. Apr 2016;103(5):504-512.
- 31. Gillis C, Li C, Lee L, et al. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. Nov 2014;121(5):937-947.
- 32. Le Roy B, Selvy M, Slim K. The concept of prehabilitation: What the surgeon needs to know? J Visc Surg. Apr 2016;153(2):109-112.
- 33. Marchand AA, Suitner M, O'Shaughnessy J, et al. Effects of a prehabilitation program on patients' recovery following spinal stenosis surgery: study protocol for a randomized controlled trial. Trials. 2015;16:483.
- 34. West MA, Loughney L, Lythgoe D, et al. Effect of prehabilitation on objectively measured physical fitness after neoadjuvant treatment in preoperative rectal cancer patients: a blinded interventional pilot study. British journal of anaesthesia. Feb 2015;114(2):244-251.
- 35. Schopfer DW, Forman DE. Cardiac Rehabilitation in Older Adults. Can J Cardiol. Mar 10 2016.
- 36. Stammers AN, Kehler DS, Afilalo J, et al. Protocol for the PREHAB study-Pre-operative Rehabilitation for reduction of Hospitalization After coronary Bypass and valvular surgery: a randomised controlled trial. BMJ Open. 2015;5(3):e007250.
- 37. Katsura M, Kuriyama A, Takeshima T, et al. Preoperative inspiratory muscle training for postoperative pulmonary complications in adults undergoing cardiac and major abdominal surgery. The Cochrane database of systematic reviews. 2015;10:Cd010356.
- 38. Sebio R, Yáñez-Brage MI, Giménez-Moolhuyzen E, et al. Impact of a Pre-Operative Pulmonary Rehabilitation Program on Functional Performance In Patients Undergoing Video-assisted Thoracic Surgery for Lung Cancer. Archivos de Bronconeumología (English Edition). 2016;52(5):231-232.
- 39. Fried LP, Tangen CM, Walston J, et al. Frailty in older adults: evidence for a phenotype. The journals of gerontology. Series A, Biological sciences and medical sciences. Mar 2001;56(3):M146-156.
- 40. Rockwood K, Mitnitski A. Frailty in relation to the accumulation of deficits. The journals of gerontology. Series A, Biological sciences and medical sciences. Jul 2007;62(7):722-727.
- 41. Hall DE, Arya S, Schmid KK, et al. Development and initial validation of the risk analysis index for measuring frailty in surgical populations. JAMA Surgery. 2016.

- 42. Guralnik JM, Simonsick EM, Ferrucci L, et al. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. Mar 1994;49(2):M85-94.
- 43. Laboratories ATSCoPSfCPF. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. Jul 1 2002;166(1):111-117.
- 44. Chatham K, Berrow S, Beeson C, et al. Inspiratory Pressures in Adult Cystic Fibrosis. Physiotherapy. 1994;80(11):758-752.
- 45. Malone A, Hamilton C. The Academy of Nutrition and Dietetics/the American Society for Parenteral and Enteral Nutrition consensus malnutrition characteristics: application in practice. Nutr Clin Pract. Dec 2013;28(6):639-650.
- 46. Hawthorne G, Richardson J, Osborne R. The Assessment of Quality of Life (AQoL) instrument: a psychometric measure of health-related quality of life. Qual Life Res. May 1999;8(3):209-224.
- 47. National Surgery Office. Annual Surgery Report: Department of Veterans Affairs; 2013.
- 48. Rodriguez-Manas L, Feart C, Mann G, et al. Searching for an operational definition of frailty: a Delphi method based consensus statement: the frailty operative definition-consensus conference project. The journals of gerontology. Series A, Biological sciences and medical sciences. Jan 2013;68(1):62-67.
- 49. Fried LP, Ferrucci L, Darer J, et al. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. The journals of gerontology. Series A, Biological sciences and medical sciences. Mar 2004;59(3):255-263.
- 50. Rockwood K, Mitnitski A. Frailty defined by deficit accumulation and geriatric medicine defined by frailty. Clinics in geriatric medicine. Feb 2011;27(1):17-26.
- 51. Inouye SK, Studenski S, Tinetti ME, et al. Geriatric syndromes: clinical, research, and policy implications of a core geriatric concept. J Am Geriatr Soc. May 2007;55(5):780-791.
- 52. Spruit MA, Singh SJ, Garvey C, et al. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. Oct 15 2013;188(8):e13-64.
- 53. Santa Mina D, Scheede-Bergdahl C, Gillis C, et al. Optimization of surgical outcomes with prehabilitation. Applied Physiology, Nutrition, and Metabolism. 2015/09/01 2015;40(9):966-969.
- 54. Furze G, Dumville JC, Miles JN, et al. "Prehabilitation" prior to CABG surgery improves physical functioning and depression. International journal of cardiology. Feb 6 2009;132(1):51-58.
- 55. Shakouri SK, Salekzamani Y, Taghizadieh A, et al. Effect of Respiratory Rehabilitation Before Open Cardiac Surgery on Respiratory Function: A Randomized Clinical Trial. Journal of Cardiovascular and Thoracic Research. 03/29 2015;7(1):13-17.
- 56. Rumer KK, Saraswathula A, Melcher ML. Prehabilitation in our most frail surgical patients: are wearable fitness devices the next frontier? Curr Opin Organ Transplant. Apr 2016;21(2):188-193.
- 57. Halloway S, Buchholz SW, Wilbur J, et al. Prehabilitation interventions for older adults: an integrative review. West J Nurs Res. Jan 2015;37(1):103-123.
- 58. Gill TM, Baker DI, Gottschalk M, et al. A prehabilitation program for physically frail community-living older persons. Arch Phys Med Rehabil. Mar 2003;84(3):394-404.
- 59. Theou O, Stathokostas L, Roland KP, et al. The effectiveness of exercise interventions for the management of frailty: a systematic review. J Aging Res. 2011;2011:569194.
- 60. de Labra C, Guimaraes-Pinheiro C, Maseda A, et al. Effects of physical exercise interventions in frail older adults: a systematic review of randomized controlled trials. BMC Geriatrics. 2015;15(1):1-16.
- 61. Daly J, Sindone AP, Thompson DR, et al. Barriers to participation in and adherence to cardiac rehabilitation programs: a critical literature review. Prog Cardiovasc Nurs. Winter 2002;17(1):8-17.
- 62. Jackson L, Leclerc J, Erskine Y, et al. Getting the most out of cardiac rehabilitation: a review of referral and adherence predictors. Heart. Jan 2005;91(1):10-14.
- 63. Pashikanti L, Von Ah D. Impact of early mobilization protocol on the medical-surgical inpatient

- population: an integrated review of literature. Clin Nurse Spec. Mar-Apr 2012;26(2):87-94.
- 64. Katsura M, Kuriyama A, Takeshima T, et al. Preoperative inspiratory muscle training for postoperative pulmonary complications in adults undergoing cardiac and major abdominal surgery. Cochrane Database of Systematic Reviews. 2015(10).
- 65. Abizanda P, Lopez MD, Garcia VP, et al. Effects of an Oral Nutritional Supplementation Plus Physical Exercise Intervention on the Physical Function, Nutritional Status, and Quality of Life in Frail Institutionalized Older Adults: The ACTIVNES Study. J Am Med Dir Assoc. May 1 2015;16(5):439 e439-439 e416.
- 66. Arnold M, Barbul A. Nutrition and wound healing. Plast Reconstr Surg. Jun 2006;117(7 Suppl):42S-58S.
- 67. Department of Veterans Affairs. Blueprint for Excellence. Veterans Health Administration [online] 2014. Accessed December 1, 2014.
- 68. Office of Geriatrics and Extended Care Services. About the Office of Geriatrics and Extended Care Services: Department of Veterans Affairs [online]. Dowloaded May 22, 2014.
- 69. Cahalin LP, Arena R. Novel methods of inspiratory muscle training via the Test of Incremental Respiratory Endurance (TIRE). Exerc Sport Sci Rev. Apr 2015;43(2):84-92.
- 70. Cahalin LP, Arena R, Guazzi M, et al. Inspiratory muscle training in heart disease and heart failure: a review of the literature with a focus on method of training and outcomes. Expert Rev Cardiovasc Ther. Feb 2013;11(2):161-177.
- 71. Cahalin LP, Semigran MJ, Dec GW. Inspiratory muscle training in patients with chronic heart failure awaiting cardiac transplantation: results of a pilot clinical trial. Phys Ther. Aug 1997;77(8):830-838.
- 72. Cahalin LP, Wagenaar R, Dec GW, et al. Endurance training in HF— A pilot study of the effects of cycle versus ventilatory muscle training. Circ. 2001;104(17):II-453.
- 73. Cahalin LP, Arena RA. Breathing exercises and inspiratory muscle training in heart failure. Heart Fail Clin. Jan 2015;11(1):149-172.
- 74. Hall DE, Arya S, Schmid KK, et al. Association of a frailty screening initiative with postoperative survival at 30, 180, and 365 days. JAMA Surgery. 2016.
- 75. Forman DE, Clare R, Kitzman DW, et al. Relationship of age and exercise performance in patients with heart failure: the HF-ACTION study. Am Heart J. Oct 2009;158(4 Suppl):S6-S15.
- 76. Yeh GY, McCarthy EP, Wayne PM, et al. Tai chi exercise in patients with chronic heart failure: a randomized clinical trial. Arch Intern Med. Apr 25 2011;171(8):750-757.
- 77. Lecker SH, Zavin A, Cao P, et al. Expression of the irisin precursor FNDC5 in skeletal muscle correlates with aerobic exercise performance in patients with heart failure. Circulation. Heart failure. Nov 2012;5(6):812-818.
- 78. Gill TM, Baker DI, Gottschalk M, et al. A program to prevent functional decline in physically frail, elderly persons who live at home. N Engl J Med. 2002;347.
- 79. Gill TM, Gahbauer EA, Allore HG, et al. Transitions between frailty states among community-living older persons. Arch Intern Med. 2006;166.
- 80. Gill TM, Guralnik JM, Pahor M, et al. Effect of Structured Physical Activity on Overall Burden and Transitions Between States of Major Mobility Disability in Older Persons: Secondary Analysis of a Randomized Trial. Annals of internal medicine. Dec 20 2016;165(12):833-840.
- 81. Greysen SR, Stijacic Cenzer I, Auerbach AD, et al. Functional impairment and hospital readmission in Medicare seniors. JAMA Intern Med. Apr 2015;175(4):559-565.
- 82. Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-381.
- 83. Fiatarone MA, Marks EC, Ryan ND, et al. High-intensity strength training in nonagenarians. Effects on skeletal muscle. Jama. Jun 13 1990;263(22):3029-3034.
- 84. Rockwood K, Song X, MacKnight C, et al. A global clinical measure of fitness and frailty in elderly people. CMAJ. Aug 30 2005;173(5):489-495.

- 85. Cesari M, Kritchevsky SB, Newman AB, et al. Added value of physical performance measures in predicting adverse health-related events: results from the Health, Aging And Body Composition Study. J Am Geriatr Soc. Feb 2009;57(2):251-259.
- 86. Guralnik JM, Ferrucci L, Simonsick EM, et al. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. Mar 2 1995;332(9):556-561.
- 87. Rolland Y, Lauwers-Cances V, Cesari M, et al. Physical performance measures as predictors of mortality in a cohort of community-dwelling older French women. European journal of epidemiology. 2006;21(2):113-122.
- 88. Guralnik JM. Assessment of physical performance and disability in older persons. Muscle & nerve. Supplement. 1997;5:S14-16.
- 89. Vasunilashorn S, Coppin AK, Patel KV, et al. Use of the Short Physical Performance Battery Score to Predict Loss of Ability to Walk 400 Meters: Analysis From the InCHIANTI Study. The Journals of Gerontology Series A: Biological Sciences and Medical Sciences. 2009;64A(2):223-229.
- 90. Beck FK, Rosenthal TC. Prealbumin: a marker for nutritional evaluation. Am Fam Physician. Apr 15 2002;65(8):1575-1578.
- 91. Measurement of visceral protein status in assessing protein and energy malnutrition: standard of care. Prealbumin in Nutritional Care Consensus Group. Nutrition. Mar-Apr 1995;11(2):169-171.
- 92. Detsky AS, McLaughlin JR, Baker JP, et al. What is subjective global assessment of nutritional status. J Parenteral and Enteral Nutrition. 1987;11(1):8-13.
- 93. Hawthorne G, Osborne R. Population norms and meaningful differences for the Assessment of Quality of Life (AQoL) measure. Aust N Z J Public Health. Apr 2005;29(2):136-142.
- 94. Slankamenac K, Graf R, Barkun J, et al. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. Jul 2013;258(1):1-7.
- 95. Moore CG, Carter RE, Nietert PJ, et al. Recommendations for planning pilot studies in clinical and translational research. Clinical and translational science. Oct 2011;4(5):332-337.
- 96. VanderWeele TJ. (2017). On the promotion of human flourishing. (Wachter, KW, ed.). Proceedings of the National Academy of Sciences of the United States of America. Aug 1 2017; 114 (31): 8148-8156.